CLINICAL TRIAL: NCT05963269
Title: The Effect of Computer Aided Game on the Development of Intramuscular Injection Application Skills of Nursing Students
Brief Title: The Effect of the Game on Students' Intramuscular Injection Skills
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Nehir Demirel, Lecturer, Maltepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MaltepeU_DemirelN
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Video Games; Students; Nursing; Infections; Intramuscular
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Students receiving computer game support in intramuscular injection learning (Active Comparator): After learning intramuscular injection with demonstration, a group of students reinforcing intramuscular injection training for 1 week with a computer-assisted game designed by the researcher.
  Interventions: Other: Computer assisted intramuscular learning game
- Group of students learning intramuscular injection only by demonstration (No Intervention): Group of students learning intramuscular injection by demonstration method without computer-assisted games

INTERVENTIONS:
Other: Computer assisted intramuscular learning game — It is an educational game that can only be opened from the computer, with questions and answers and cases. The game is currently under development by the developers. The researcher will be able to see how many times the students entered the game and how many points they got.
  Arms: Students receiving computer game support in intramuscular injection learning

SUMMARY:
Today, error rates increase in intramuscular (IM) drug administrations, which are frequently applied in clinical settings, due to many factors such as the increase in the number of students in nursing education, the low number of educators, insufficient clinical space and insufficient laboratory environments. This situation makes it inevitable to use different teaching methods in nursing education, especially in the acquisition and development of psychomotor skills. Games, which are a type of virtual simulation methods; It is defined as a pedagogical tool that offers the student the widest possible learning opportunity, interesting, interactive media, and a teaching beyond entertainment. It is very important to acquire the necessary knowledge and skills in the management of intramuscular drug administration, which will constitute the majority of postgraduate applications of nursing students, by using today's technologies during their student life. Another factor that is effective in psychomotor skill learning is; students' anxiety level. Nursing students may experience anxiety while using the new technique, which negatively affects the learning process of the student. One of the reasons for the anxiety experienced by the students is that they have not reached enough professional knowledge and skills. It is observed that this level of anxiety increases especially in psychomotor skills. In the exams conducted for the evaluation of laboratory practices in nursing education, the student demonstrates the skills learned during the term. The level of anxiety he feels during this practice may also affect his performance. The general result of studies examining the relationship between test anxiety and academic performance is that there is a negative relationship between test anxiety and academic success. For this reason, it is very important to control students' anxiety. Although the level of state anxiety increases from time to time, especially in the trainings carried out with simulation, it is one of the training methods that increases the self-confidence of the students by reducing their anxiety in the future. Based on these reasons, this research; The aim of this study was to evaluate the effect of computer-assisted game on success and anxiety level in the development of intramuscular injection application skills in nursing education.

ELIGIBILITY:
Inclusion Criteria:

* Being a first year nursing student
* To be taking the basics of nursing course for the first time
* To have at least 50 points from the IM Injection Information Form

Exclusion Criteria:

* Graduated from Health Vocational High School
* Having a communication problem related to vision and hearing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-08-28 (Estimated); Study Completion 2023-09-29 (Estimated)

PRIMARY OUTCOMES:
Computer-assisted games change students' knowledge about IM injection. | 2 week
  1 week after playing the game, the level of knowledge will be evaluated by an independent observer with a practice exam.

CONTACTS AND LOCATIONS:
Locations (1):
- Maltepe University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The collected data will not be shared with any institution or legal person.